CLINICAL TRIAL: NCT04754282
Title: Impact of a Cross-legged Versus Traditional Sitting Position for the Success of an Epidural Analgesia Catheter Placement During Labor
Brief Title: Cross-legged Versus Traditional Sitting Position for the Success of Epidural Analgesia During Labor
Acronym: IP3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP201193; 2020-A02267-32 (Other: ID-RCB Number)
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Epidural Analgesia for Labour and Delivery
Keywords: Epidural anesthesia; Sitting position; Cross-legged position; Labour; Pain; Obstetric
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional sitting position (Active Comparator): Expecting women are positioned in a traditional sitting position for epidural analgesia catheter placement during labour.
  Interventions: Other: Position of labouring women for epidural analgesia catheter placement : Traditional Sitting Position (TSP)
- Cross-legged sitting position (Experimental): Expecting women are positioned in a crosse-legged sitting position for epidural analgesia catheter placement during labour.
  Interventions: Other: Position of labouring women for epidural analgesia catheter placement : Cross-legged Sitting Position (CSP)

INTERVENTIONS:
Other: Position of labouring women for epidural analgesia catheter placement : Traditional Sitting Position (TSP) — Labouring women admitted to the delivery room of Necker Enfants Malades hospital, requesting an epidural analgesia for labour, and willing to participate in our study will be randomized in the Traditional Sitting Position (TSP) group on odd days or in the Cross-legged Sitting Position (CSP) group on even days.
  Patients in the TSP group seat on the edge of the bed, their feet laid on a support set next to the bed. Patients in the CSP group also seat on the edge the bed, but in a so-called "tailor" position, their knees bent, their hips flexed and in abduction, their feet under each contralateral thigh.
  The epidural catheter will be placed according to standard local practice in either of the groups.
  Other Names: Traditional Sitting Position (TSP)
  Arms: Traditional sitting position
Other: Position of labouring women for epidural analgesia catheter placement : Cross-legged Sitting Position (CSP) — Labouring women admitted to the delivery room of Necker Enfants Malades hospital, requesting an epidural analgesia for labour, and willing to participate in our study will be randomized in the Traditional Sitting Position (TSP) group on odd days or in the Cross-legged Sitting Position (CSP) group on even days.
  Patients in the TSP group seat on the edge of the bed, their feet laid on a support set next to the bed. Patients in the CSP group also seat on the edge the bed, but in a so-called "tailor" position, their knees bent, their hips flexed and in abduction, their feet under each contralateral thigh.
  The epidural catheter will be placed according to standard local practice in either of the groups.
  Other Names: Cross-legged Sitting Position (CSP)
  Arms: Cross-legged sitting position

SUMMARY:
The success of an epidural analgesia catheter placement depends on the parturient position. A poor posture can increase the number of punctures, patient discomfort, and risk of complications. An adequate position reverses lumbar lordosis, facilitating the access to the intervertebral space. In most cases, insertion of the epidural analgesia catheter is performed in sitting position or in lateral decubitus, the choice being generally guided by the preference of the anesthetist.

According to anesthetists' experience in the obstetrical anesthesia unit at Necker-Enfants Malades hospital, a cross-legged sitting position is comfortable for parturients, restricts interfering movements during the procedure, and provides adequate widening of interspinous spaces. This position results in knees and hips flexion, tilting the pelvis backward and opening the interspinous spaces, while limiting muscular strain to maintain the position. However, literature on this matter is scarce.

The aim of this study is to prove the superiority of the cross-legged position for successful placement of the epidural analgesia catheter at the first puncture without needle reorientation compared to a traditional sitting position on the edge of the bed.

DETAILED DESCRIPTION:
Labour pain is one of the most intense pain known. To relieve this pain, epidural analgesia is both the most effective and the safest technique. An epidural analgesia catheter also allows for anesthesia in the event of the need for instrumental extraction or emergency caesarean section; it is thus recommended by learned societies.

The 2016 national perinatal survey conducted by the National Institute of Health and Medical Research (INSERM) and the Directorate of Research, Studies, Evaluation and Statistics (DREES) in France revealed that more than 80% of women had chosen to benefit from an epidural analgesia during labour. The first puncture failure rate ranges from 3% to almost 40% depending on the study. Identified factors for difficult epidural analgesia catheter placement were: non-palpable spinous processes, obesity, spine deformity, inability for the patient to maintain an adequate position and poor experience of the operator.

The success of an epidural analgesia catheter placement depends on the parturient position. A poor posture can increase the number of punctures, patient discomfort, and risk of complications. An adequate position reverses lumbar lordosis, facilitating the access to the intervertebral space. Different positions have been described: the lateral decubitus, the traditional sitting position, and its variants such as the squatting position, the "hamstring stretch" position, the "pendant position" (with a bilateral axillary support) and more recently the cross-legged position. In most cases, insertion of the epidural analgesia catheter is performed in sitting position or in lateral decubitus, the choice being generally guided by the preference of the anesthetist.

According to anesthetists' experience in the obstetrical anesthesia unit at Necker-Enfants Malades hospital, a cross-legged sitting position is comfortable for parturients, restricts interfering movements during the procedure, and provides adequate widening of interspinous spaces. This position results in knees and hips flexion, tilting the pelvis backward and opening the interspinous spaces, while limiting muscular strain to maintain the position. However, literature on this matter is scarce.

The aim of this study is to prove the superiority of the cross-legged position for successful placement of the epidural analgesia catheter at the first puncture without needle reorientation compared to a traditional sitting position on the edge of the bed.

ELIGIBILITY:
Inclusion Criteria:

* Adult women admitted to the delivery room and requesting an epidural analgesia during labour
* Written informed consent
* French speaking patient

Exclusion Criteria:

* Patient with a contraindication to neuraxial analgesia
* Impossibility for the patient to seat in a cross-legged position
* No health insurance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 457 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-03-26 (Actual); Study Completion 2022-03-26 (Actual)

PRIMARY OUTCOMES:
Epidural analgesia success rate | 20 minutes
  Percentage of epidural analgesia catheter placement success at first puncture without needle reorientation

SECONDARY OUTCOMES:
Patient's comfort | 20 minutes
  Visual Analog Scale (VAS) comfort score (0 (maximum discomfort) to 10 (maximum comfort)) of parturients during the epidural analgesia catheter placement
Patient's pain | 20 minutes
  VAS pain score (0 (no pain) to 10 (worst imaginable pain)) of parturients during the epidural analgesia catheter placement
Epidural analgesia success rate in obese patients | 20 minutes
  Percentage of epidural analgesia catheter placement success at first puncture without needle reorientation in the subpopulation of obese patients
Successful rate of epidural analgesia catheter placement by residents | 20 minutes
  Percentage of epidural analgesia catheter placement success at first puncture without needle reorientation for epidurals placed by anaesthetist residents
Operator satisfaction | 20 minutes
  VAS satisfaction score (0 (maximum dissatisfaction) to 10 (maximum satisfaction)) of the operator in relation to the parturient's position during the procedure
Adverse event occurrence rate | 20 minutes
  Percentage of intra-vascular catheter position, dura-mater puncture, paraesthesia, hypotension after epidural analgesia initiation

CONTACTS AND LOCATIONS:
Overall Officials: Hawa KEITA-MEYER, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Kevin SEREY, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serey K, Osse L, Repesse X, Babou J, Banna L, Ayoub M, Elseblani R, Brebion M, Keita H. Cross-legged position versus traditional sitting position for epidural catheter insertion for labor analgesia: a non-randomized prospective study. Int J Obstet Anesth. 2024 Feb;57:103938. doi: 10.1016/j.ijoa.2023.103938. Epub 2023 Oct 11. No abstract available. PMID 37891125